CLINICAL TRIAL: NCT00676156
Title: A Pilot Trial to Study the Pharmacokinetics of Oral Lipoic Acid (LA) and Immunological Effects of LA in Multiple Sclerosis
Brief Title: A Study of the Pharmacokinetics and Immunologic Effects of Lipoic Acid in Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Vijayshree Yadav, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB00001305; NCCAM 1K23 AT003258-01
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; lipoic acid; LA; pharmacokinetics; immunological effects
MeSH Terms: conditions — Multiple Sclerosis | interventions — Thioctic Acid; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): This arm involves a 1-day pharmacokinetics study of three different formulations of oral lipoic acid.
  Interventions: Drug: oral lipoic acid (LA)
- B (Active Comparator): This arm will examine the pharmacokinetics of LA with and without fish oil supplement in a cross over design.
  Interventions: Drug: lipoic acid (LA) with fish oil and LA without fish oil
- C (Active Comparator): This arm will include the study of a single dose of R enantiomer lipoic acid.
  Interventions: Drug: R lipoic acid

INTERVENTIONS:
Drug: oral lipoic acid (LA) — A single 1200 mg dose of oral LA will be administered.
  Arms: A
Drug: lipoic acid (LA) with fish oil and LA without fish oil — Subjects will be randomized to receive either 1 dose of 1200 mg LA with fish oil and then will be crossed-over to receive 1 dose of 1200 LA without fish oil. There will be a 1-week wash out period between the cross over.
  Arms: B
Drug: R lipoic acid — A single oral dose of 1200mg R enantiomer LA will be administered.
  Arms: C

SUMMARY:
The purpose of this study is to learn about an investigational drug known as oral lipoic acid (LA) that may help treat multiple sclerosis. This study will measure how a person's body absorbs and breaks down the drug (pharmacokinetics) and will compare four different forms of the drug from four different manufacturers as well as LA in conjunction with fish oil.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a common, often disabling inflammatory disease of the central nervous system (CNS). Present treatments for MS are only partially effective, available only in injectable forms, have significant side effects and are very costly. Developing more effective and better-tolerated treatments of MS thus remains an important goal for the improvement of the care of MS. Lipoic acid (LA) is an antioxidant that is widely available as a dietary supplement.

The primary outcome of this study is to determine the pharmacokinetics of oral LA 1200 mg to see if we can identify factors affecting the bioavailability of LA. We will also study the salivary concentrations of oral LA and its correlation with the serum LA concentrations. We will also study the effects of LA on the immunological markers after four hours of administration.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS by McDonald's or Poser's criteria
* EDSS ≤ 7.5
* Age 18 to 80

Exclusion Criteria:

* No clinically significant MS exacerbation within 30 days of the screening
* No systemically administered corticosteroids within 30 days of study entry
* Patient not pregnant or breast feeding
* No LA in previous 2 weeks
* Not on anti-coagulants such as heparin, coumadin, or aspirin during study
* No other significant health problem (e.g. active coronary heart disease, liver disease, pulmonary disease, diabetes mellitus) that might increase risk of patient experiencing adverse events
* Inability to give informed consent
* Any condition which would make the patient, in the opinion of the investigator, unsuitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetics of orally administered LA 1200 mg. This will assess the variability in bioavailability of LA and the feasibility of conducting a more focused PK assessment in future studies with LA. | November 2008

SECONDARY OUTCOMES:
To study salivary LA concentrations corresponding to the serum levels. | November 2008

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University Multiple Sclerosis Dept., Portland, Oregon, United States